CLINICAL TRIAL: NCT00755872
Title: Influence of a High-fat Meal on the Bioavailability of a Two Different Formulations of Risedronate
Brief Title: Assess the Influence of a High-fat Meal on the Relative Bioavailability Of Two Formulations of Risedronate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2007120
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Bioavailability
MeSH Terms: interventions — Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Treatment A (35 mg DR Fasted): One risedronate tablet (35 mg DR) taken following an overnight (10-hour) fast, followed by a 4-hour fast.
  Interventions: Drug: Risedronate
- 2 (Experimental): Treatment B (35 mg DR Fed): One risedronate tablet (35 mg DR) taken following an overnight (10-hour) fast, within 5 minutes after ingesting a high-fat meal.
  Interventions: Drug: Risedronate
- 3 (Experimental): Treatment C (35 mg IR Fasted): One risedronate tablet (35 mg IR) taken following an overnight (10-hour) fast, followed by a 4-hour fast.
  Interventions: Drug: Risedronate
- 4 (Experimental): Treatment D (35 mg IR Per-label): One risedronate tablet (35 mg IR) taken following an overnight (10-hour) fast, 30 minutes before ingesting a high-fat meal.
  Interventions: Drug: Risedronate

INTERVENTIONS:
Drug: Risedronate — Treatment A (35 mg DR Fasted): One risedronate tablet (35 mg DR) taken following an overnight (10-hour) fast, followed by a 4-hour fast.
  Arms: 1
Drug: Risedronate — Treatment B (35 mg DR Fed): One risedronate tablet (35 mg DR) taken following an overnight (10-hour) fast, within 5 minutes after ingesting a high-fat meal.
  Arms: 2
Drug: Risedronate — Treatment C (35 mg IR Fasted): One risedronate tablet (35 mg IR) taken following an overnight (10-hour) fast, followed by a 4-hour fast.
  Arms: 3
Drug: Risedronate — Treatment D (35 mg IR Per-label): One risedronate tablet (35 mg IR) taken following an overnight (10-hour) fast, 30 minutes before ingesting a high-fat meal.
  Arms: 4

SUMMARY:
This is a randomized, open-label, multi-center, 4-treatment, 4-period crossover study. Approximately 72 healthy, surgically sterile or postmenopausal subjects will be enrolled and have urine collected over 72 hours following administration of risedronate for all 4 treatment periods).

ELIGIBILITY:
Inclusion Criteria:

* Females 40 - 70 years at time of first dose
* BMI less than or equal to 32 kg/square meter
* Non-lactating and either surgically sterile or postmenopausal

Exclusion Criteria:

* Clinically significant uncontrolled cardiovascular, hepatic, renal, or thyroid disease
* Had a major surgical operation requiring inpatient hospitalization within 1 month prior to screening or plans to have a major surgical operation during the course of the study
* A history of cancer within the past 5 years, except for basal cell carcinoma with documentation of a 6-month remission at screening. Subjects with a more recent history of successfully treated cervical carcinoma in situ will not be excluded, provided there is documentation of a 12-month remission
* Any disease or surgery known to alter normal gastrointestinal structure or function
* A history of gastrointestinal disease (peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease, irritable bowel syndrome, or moderate to severe gastro-esophageal reflux disease that requires prescription or frequent [> 3 times/week] nonprescription medicinal intervention [eg, antacids])
* A history of gastrointestinal surgery, with the exception of appendectomy and hernia repair that did not require bowel resection (subjects who have undergone appendectomy or hernia repair within the 12 months prior to screening will be excluded from the study)
* Acute gastritis, diarrhea or constipation within the 14-day period prior to the predicted first dosing day. If screening occurs >14 days before the first dosing day, subjects will be re-evaluated for eligibility at admission. Diarrhea will be defined as the passage of liquid feces and/or a stool frequency of greater than 3 times per day. Constipation will be defined as having less than 3 bowel movements per week or as having fewer bowel movements than is usual for the subject

Exclusion at Admission:

* Any significant change from screening which in the investigator's opinion would impact safety of subject or interfere with the evaluation of the study drug.
* Had any acute illness within the past 2 weeks.
* Consumed alcohol, grapefruit or grapefruit juice, orange juice, chocolate, or caffeine within 72 hours of dosing.
* Used a bisphosphonate since screening.
* Reported exposure to any known enzyme inducer or inhibitor, transport induceror inhibitor or nonmedical enzyme-inducers such as paint solvents or pesticides since screening.
* A positive pregnancy test.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Assess the relative bioavailability of the 35 mg DR risedronate tablet administered immediately after a high-fat meal compared to the 35 mg IR risedronate tablet administered 30 minutes prior to a high-fat meal. | 4 Days

SECONDARY OUTCOMES:
Assess the relative bioavailability of a 35 mg DR risedronate tablet administered immediately after a high-fat meal compared to the same 35 mg DR risedronate tablet administered under fasted conditions. | 4 Days

CONTACTS AND LOCATIONS:
Overall Officials: William S Aronstein, MD, PhD, Study Director — Procter and Gamble
Locations (3):
- United States (3):
  - Research Site, Fort Myers, Florida
  - Research Site, Miramar, Florida
  - Research Site, Austin, Texas